CLINICAL TRIAL: NCT02485366
Title: Rejuvenated, Washed Packed Red Blood Cells in Pediatric Cardiac Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Product unavailability
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00021487
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Heart Defects, Congenital
Keywords: Rejuvenated packed red blood cells
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rejuvenated PRBCs (Experimental): The investigators will restore important energy molecules in stored red blood cells before they are transfused, with a rejuvenating solution (Rejuvesol).
  Interventions: Drug: Rejuvesol; Procedure: Cardiac surgery

INTERVENTIONS:
Drug: Rejuvesol — Blood transfused during surgery will be treated with Rejuvesol.
Procedure: Cardiac surgery — The study interventions will take place during a routine admission for pediatric open heart surgery. The anesthetic technique for subjects undergoing cardiac surgery is standard care and the research study interventions will not change these practices in any way.

SUMMARY:
Blood transfusion is nearly always needed during open heart surgery in children less than 15 kg (35 pounds). The purpose of the red blood cells in the blood is to deliver oxygen to the organs and tissues of the body. Stored blood undergoes some changes that may make it less effective in achieving this goal. The purpose of this study is to see if restoring important energy molecules (ATP and 2,3,DPG) in stored red blood cells before they are transfused, with a rejuvenating solution (Rejuvesol), offers any advantages to children over standard blood transfusion. This is a Food and Drug Administration (FDA) approved process that is described by the American Association of Blood Banks for prolonging blood storage but not used for everyday transfusions. The investigators want to use this process to improve blood transfused to children undergoing heart surgery.

Although Rejuvesol has been previously approved by the FDA, it is not routinely used to prepare standard blood transfusions to children undergoing surgery. Use of Rejuvesol in this study is considered investigational. This is a pilot study and data will be collected for future protocol development.

ELIGIBILITY:
Inclusion Criteria:

* children greater than 2.5 kg and less than 15kg (i.e. requiring blood for CPB prime)
* children undergoing cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* refusal of blood products
* end-stage renal disease
* planned avoidance of CPB
* use of non- heparin anticoagulants
* participation in an experimental drug or device protocol within 30 days
* existing hemoglobinopathy
* allergy requiring washed RBCs
* immunocompromise requiring special blood product treatment.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in tissue oxygenation/perfusion during cardiac surgery, measured by whole blood lactate concentration | End of Surgery
Change in ischemic organ injury during cardiac surgery, measured by urinary neutrophil gelatinase associated lipocalin (NGAL) | 2 hours
Change in hemolysis during cardiac surgery, as measured by plasma free hemoglobin levels | end of bypass

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lodge, MD, Principal Investigator — Duke University
Locations (1):
- Duke Univerisity Medical Center, Durham, North Carolina, United States